CLINICAL TRIAL: NCT06521749
Title: Evaluating the Use of the Universal Stylet Bougie (USB) on Successful Intubation on the First Attempt Among Patients with Cervical Spine Immobilization by Using a Rigid Collar.
Brief Title: Universal Stylet Bougie in Patients with Cervical Neck Immobilization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Assistant lecturer, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PT(823)
Record Dates: First submitted 2024-07-21; First posted 2024-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Intubating Condition
Keywords: USB, cervical immobilization, rigid collar

STUDY DESIGN:
Intervention Model Description: Patients will be allocated, according to the study group into:
  1. Bougie Group: (Group A) Endotracheal intubation will be attempted using the video laryngoscope and the USB device will be used as a bougie.
  2. Stylet Group: ( Group B) Endotracheal intubation will be attempted using the video laryngoscope and using the USB device as a stylet.
  3. Control Group: (Group C) Intubation of the trachea with an endotracheal tube will be attempted by using only the video laryngoscopy.
Who Masked: Participant, Outcomes Assessor
Masking Description: the investigator responsible for data collection and the patients participating in the study will not be aware of the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the Bougie group (group A) (Active Comparator): Endotracheal intubation will be attempted using the video laryngoscope and the USB device will be used as a bougie.
  Interventions: Device: USB as a bougie
- the stylet group ( B group) (Active Comparator): Endotracheal intubation will be attempted using the video laryngoscope and using the USB device as a stylet.
  Interventions: Device: USB as a stylet
- the control group (C group) (No Intervention): Intubation of the trachea with an endotracheal tube will be attempted by using only the video laryngoscopy.

INTERVENTIONS:
Device: USB as a stylet — USB used as a bougie
  Arms: the stylet group ( B group)
Device: USB as a bougie — USB used as a bougie
  Arms: the Bougie group (group A)

SUMMARY:
In patients with cervical spine injury, securing the airway while adequately immobilizing the cervical spine to avoid secondary neurological damage is very challenging. Although awake fiber-optic intubation is the most reliable method in patients with cervical trauma, it has some limitations such as lack of availability, need for expertise in the use, difficulty with non-cooperative patients, or presence of blood or secretions in the airway. Two devices are commonly used to facilitate tracheal intubation: a stylet or a tracheal tube introducer ("bougie").

DETAILED DESCRIPTION:
The Universal Stylet Bougie, or USB™, represents a significant advance in the design and development of tracheal introducers (bougies) and stylets. Traditionally, the design requirements of styles and bougies have always been considered incompatible. A stylet requires sufficient rigidity to allow the tracheal tube to be manipulated to a variety of angles, whereas a bougie needs to be flexible enough to allow positive tracheal ring feedback to allow correct placement.

The unique design of the USB™ means the device can be used as a stylet or as a bougie. It consists of two metals inserted on both sides and a flexible middle section. The USB can easily be manipulated to a variety of angles when used as a stylet, yet has the flexibility when used as a bougie. In addition, the hexagonal shape provides less contact with the inner surface of the tracheal tube, providing particularly easy insertion and removal.

In this study we are simulating a difficult intubating condition by limiting the cervical neck extension through applying a rigid neck collar. Subsequently, we will assess whether using the USB device could improve the successful rate of intubation in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. ASA (American society of Anesthesiologists) physical status 1-2.
2. Age 18- 60 years old of both sexes.
3. Patients undergoing elective surgery under general anesthesia and tracheal intubation.

Exclusion Criteria:

1. Age < 18 years and ≥ 60 years
2. Pregnancy
3. Patients with BMI >35 kg m-2
4. Emergency surgery or full stomach
5. Patients with suspected difficult airway {e.g., high neck circumference, airway masses, mouth scars, neck scars, or history of snoring).
6. Patients with cervical spine pathology
7. Patients with any cardiac disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Time required for intubation. | 30 seconds - 2 minutes

SECONDARY OUTCOMES:
number of attempts | 30 seconds to 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Moshira Amer, M.D., Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available upon request from the principal investigator.

REFERENCES:
- [Background] Maremanda KR, Jayaram K, Durga P. Comparison of Intubation Conditions Between Airtraq, McGrath Video Laryngoscopes, and Macintosh Under Conditions of Simulated Trauma Airway and Rapid Sequence Induction Intubation. J Emerg Med. 2023 Mar;64(3):271-281. doi: 10.1016/j.jemermed.2022.12.014. Epub 2023 Mar 2. PMID 36868945
- [Background] Karlsen KAH, Gisvold SE, Nordseth T, Fasting S. Incidence, causes, and management of failed awake fibreoptic intubation-A retrospective study of 833 procedures. Acta Anaesthesiol Scand. 2023 Nov;67(10):1341-1347. doi: 10.1111/aas.14313. Epub 2023 Aug 16. PMID 37587618
- [Background] Kuo YM, Lai HY, Tan EC, Li YS, Chiang TY, Huang SS, Huang WC, Chu YC. Cervical spine immobilization does not interfere with nasotracheal intubation performed using GlideScope videolaryngoscopy: a randomized equivalence trial. Sci Rep. 2022 Mar 8;12(1):4041. doi: 10.1038/s41598-022-08035-0. PMID 35260735